CLINICAL TRIAL: NCT05861349
Title: Utility of the Measurement of Median Nerve Stenosis for Diagnosis of Carpal Tunnel Syndrome
Brief Title: Median Nerve Stenosis in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Jakub Antczak (Other)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Organization: Jagiellonian University (Other)
Other Study IDs: JagiellonianU71
Record Dates: First submitted 2023-05-03; First posted 2023-05-16 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; ultrasound; nerve compression
MeSH Terms: conditions — Carpal Tunnel Syndrome; Neuroma | interventions — Nerve Conduction Studies; Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CTS: Patients referred to the Electromyographic Laboratory of the Department of Neurology at the Jagiellonian University Medical College, Cracow, Poland with symptoms suggestive of CTS (numbness of the hand, present or accentuated in the night, reduced hand dexterity) with CTS confirmed in NCS or US.
  Interventions: Diagnostic Test: Nerve conduction study; Diagnostic Test: Ultrasound
- Healthy controls: Subjects referred to the Electromyographic Laboratory of the Department of Neurology at the Jagiellonian University Medical College, Cracow, Poland for investigation towards tetany, with no or only weak signs of tetany in electromyography.
  Interventions: Diagnostic Test: Nerve conduction study; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Nerve conduction study — Nerve conduction study of median and ulnar nerve together with sensory comparative methods on the affected side (sides).
Diagnostic Test: Ultrasound — Ultrasound of the median nerve on the affected side (sides).

SUMMARY:
The goal of this observational study is to test the new kind of ultrasound-based measurements in patients with carpal tunnel syndrome. The main questions it aims to answer are:

* Do the measurements of the size of the median nerve at the point where it is maximally compressed accurately diagnose carpal tunnel syndrome?
* May these measurements accurately tell how severe is the carpal tunnel syndrome?

Participants will be asked to:

* Undergo conduction studies of median and ulnar nerve.
* Undergo ultrasound of the median nerve.
* Fill out the Boston carpal tunnel questionnaire and a demographic questionnaire.

Researchers will compare the group of patients with carpal tunnel syndrome with healthy volunteers to see if respective measurements differ significantly between groups.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compression neuropathy. CTS results from the compression of the median nerve in the carpal tunnel. The main symptoms include pain and other unpleasant sensations in hand and wrist. In more advanced stage, weakness and wasting of the thenar and other muscles innervated by median nerve occurs, which may lead to permanent impairment of manual performance. Nerve conduction studies (NCS) remain the method of choice in diagnosing CTS. However ultrasonography (US) is increasingly used along with or instead of NCS. Most frequently, the increase of the cross-sectional area of the median nerve at the inlet to the carpal tunnel is regarded as the marker of CTS. A number of other measurements such as median nerve mobility, volar bulging of flexor retinaculum and others were also studied to increase diagnostic sensitivity and specificity. In this study the investigators aim to assess the utility of measurements made at the point of the maximal stenosis of the median nerve in the tunnel to diagnose CTS. So far, there were only few studies, which visualized the maximal nerve stenosis, which is the essential pathological feature of CTS. In general, the group of patients with CTS and controls will undergo NCS of symptomatic median and ipsilateral ulnar nerves and US of the symptomatic median nerve with measurements of the cross-sectional area, diameter and echogenicity at various points, including the point of the maximal stenosis. The location of the maximal stenosis with respect to external (distal crease) and internal (wrist and hand bones and thenar musculature) will also be evaluated. Subjects will also be asked to fill out the Boston Carpal Tunnel Questionnaire (BCTQ) and a demographic questionnaire. US measurements will be compared between patients and healthy volunteers. US measurements, especially those made at the point of stenosis will be correlated among patients with clinical severity of CTS, reflected by the score in BCTQ and with the grade of electrophysiological severity as introduced by Padua et al. [1].

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of CTS
* Electrophysiologic and/or ultrasonographic confirmation of CTS diagnosis

Exclusion Criteria:

* Psychiatric or cognitive conditions with may disturb participation in the study
* Peripheral neuropathy in history
* Fractures and severe trauma in the area of the wrist in history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the patients referred to the EMG Laboratory of the Department of Neurology at Jagiellonian University Medical College for verification of clinical diagnosis of CTS. After NCS and/or US confirms the CTS, the patient will be asked if she/he would like to take part in the study. Healthy controls will be recruited from the patients referred for verification of clinical diagnosis of tetany, after EMG reveals weak tetany or does not confirm it.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Difference in the diameter of median nerve in the site of its maximal compression | Through study completion, an average of 1 year.
  Difference in the diameter of median nerve in the site of its maximal compression between patients with CTS and healthy controls.
Difference in the cross-sectional area of median nerve in the site of its maximal compression | Through study completion, an average of 1 year.
  Difference in the cross-sectional area of median nerve in the site of its maximal compression between patients with CTS and healthy controls.
Difference in the echogenicity of median nerve in the site of its maximal compression | Through study completion, an average of 1 year.
  Difference in the echogenicity of median nerve in the site of its maximal compression between patients with CTS and healthy controls.

SECONDARY OUTCOMES:
Correlation of the diameter of median nerve in the site of its maximal compression with BCTQ score | Through study completion, an average of 1 year.
  Correlation of the diameter of median nerve in the site of its maximal compression with BCTQ score in patients with CTS.
Correlation of the cross-sectional area of median nerve in the site of its maximal compression with BCTQ score | Through study completion, an average of 1 year.
  Correlation of the cross-sectional area of median nerve in the site of its maximal compression with BCTQ score in patients with CTS.
Correlation of echogenicity of median nerve in the site of its maximal compression with BCTQ score | Through study completion, an average of 1 year.
  Correlation of echogenicity of median nerve in the site of its maximal compression with BCTQ score in patients with CTS.
Correlation of the diameter of median nerve in the site of its maximal compression with CTS electrophysiological severity grade | Through study completion, an average of 1 year.
  Correlation of the diameter of median nerve in the site of its maximal compression with CTS electrophysiological severity grade in patients with CTS.
Correlation of the cross-sectional area of median nerve in the site of its maximal compression with CTS electrophysiological severity grade | Through study completion, an average of 1 year.
  Correlation of the cross-sectional area of median nerve in the site of its maximal compression with CTS electrophysiological severity grade in patients with CTS.
Correlation of echogenicity of median nerve in the site of its maximal compression with CTS electrophysiological severity grade | Through study completion, an average of 1 year.
  Correlation of echogenicity of median nerve in the site of its maximal compression with CTS electrophysiological severity grade in patients with CTS.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka M Fryźlewicz, MD, Study Director — Jagiellonian University Medical College, Department of Neurology; Gabriela G Rusin, MD, Study Chair — Jagiellonian University Medical College, Department of Neurology
Locations (1):
- Jagiellonian University Medical College, Department of Neurology, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
After completing the study, the age and gender of participants as well as the scores of BCTQ, the results of NCS and the US images in .jpg and .dicom will be available to other researchers on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the study results will be published.
Access Criteria: On request sent by e-mail to jakub.antczak@uj.edu.pl

REFERENCES:
- [Background] Padua L, LoMonaco M, Gregori B, Valente EM, Padua R, Tonali P. Neurophysiological classification and sensitivity in 500 carpal tunnel syndrome hands. Acta Neurol Scand. 1997 Oct;96(4):211-7. doi: 10.1111/j.1600-0404.1997.tb00271.x. PMID 9325471